CLINICAL TRIAL: NCT06960109
Title: Effect of the Mindfulness-Based Stress Reduction Program on Prenatal Attachment, Distress and Anxiety Levels in Pregnant Women With Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AEŞH-EK1-2023-267
Record Dates: First submitted 2025-04-11; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Gestational Diabetes Mellitus (GDM); Mindfulness; Prenatal Attachment; Distress; Anxiety
Keywords: Gestational Diabetes Mellitus; Mindfulness; Prenatal attachment; Prenatal Distress; Anxiety; Midwifery
MeSH Terms: conditions — Diabetes, Gestational; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: In a randomized controlled trial, pregnant women with gestational diabetes were divided into two groups: 25 intervention groups and 25 controls. The intervention group received the Mindfulness-Based Stress Reduction Program for Pregnant Women with Gestational Diabetes for 4 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: Mindfulness-Based Stress Reduction Program (Active Comparator): A Mindfulness-Based Stress Reduction Program for Pregnant Women with Gestational Diabetes was applied to 25 pregnant women with gestational diabetes in the intervention group, 2 sessions per week for 4 weeks, for a total of 8 sessions.
  Interventions: Behavioral: A Mindfulness-Based Stress Reduction Program for Pregnant Women with Gestational Diabetes
- Routine Care (Control Group) (No Intervention): 25 pregnant women with gestational diabetes in the control group received only routine prenatal care without any additional intervention.

INTERVENTIONS:
Behavioral: A Mindfulness-Based Stress Reduction Program for Pregnant Women with Gestational Diabetes — The Gestational diabetes mellitus(GDM) pregnant women in the intervention group who agreed to participate in the study and completed the pre-test were invited to the WhatsApp group created by the researcher. 3 separate groups were created with a maximum of 11 participants in each group. The days (for example; Group 1: Tuesday, Saturday) on which the program, which will continue for 4 weeks, will be implemented were determined, considering the participants in each group and the times they were available. For each group, the conscious awareness-based stress reduction program for pregnant women with GDM; For 4 weeks, there were 8 sessions, 2 sessions per week, with each session varying in duration, for an average of 45-60 minutes. The program was carried out using the Google Meet application created online by the researcher, and the connection details were shared with the participants via WhatsApp groups. In the implementation of the mindfulness-based stress reduction program for pregnant
  Arms: Intervention group: Mindfulness-Based Stress Reduction Program

SUMMARY:
This randomized controlled study aims to evaluate the potential effects of a mindfulness-based stress reduction (MBSR) program on prenatal attachment, distress, and anxiety levels among pregnant women diagnosed with gestational diabetes mellitus (GDM). The study was conducted at Ankara Etlik City Hospital between October 2023 and 2024, and included 50 pregnant women with GDM, randomly assigned to an intervention group (n=25) or a control group (n=25). The MBSR program was implemented online for the intervention group, delivered in 8 sessions over 4 weeks.

DETAILED DESCRIPTION:
DATA COLLECTION Data were collected by the principal investigator from pregnant women who applied to the Perinatology Clinic and met the inclusion criteria. The study adhered to the principles of the Declaration of Helsinki. Written informed consent was obtained from each participant. After the purpose and importance of the study were explained to eligible and voluntarily participating individuals, pre-test questionnaire forms were administered face-to-face. The forms were completed using the self-report method. In shared rooms, participants were directed to a quiet room to ensure privacy. Any questions raised by the participants were answered before and during the data collection process. Completion of the forms took approximately 10-15 minutes per participant.

To collect post-test data, an online survey was created using Google Forms. The link was distributed via WhatsApp groups established in the fourth week after the training. Participants in these groups completed the forms using the shared link.

MINDFULNESS-BASED STRESS REDUCTION PROGRAM FOR PREGNANT WOMEN WITH GESTATIONAL DIABETES MELLITUS

Preliminary Preparation Prior to initiating the intervention, the principal investigator attended an eight-week Mindfulness-Based Stress Reduction (MBSR) Program organized by the Mindfulness Institute (14.02.2023-04.04.2023), led by Prof. Dr. Zümra Atalay.

Preparation of Training Content The training content of the MBSR program tailored for pregnant women with gestational diabetes was developed based on a literature review and the training received. Expert opinions were obtained from three professionals in obstetrics, gynecology, and midwifery to assess the content's relevance and applicability. Revisions were made according to their feedback, and the finalized version was completed.

Implementation of the Program Participants in the intervention group who completed the pre-test and agreed to join the program were included in WhatsApp groups created by the principal investigator. Three separate groups were formed, each comprising a maximum of 11 participants. Group-specific training schedules (e.g., Group 1: Tuesdays and Saturdays) were arranged according to participant availability. The MBSR program was conducted over four weeks, consisting of eight sessions (two sessions per week), each lasting approximately 45-60 minutes.

Sessions were conducted via Google Meet. The training incorporated PowerPoint presentations, verbal instruction, Q&A, and mindfulness exercises (e.g., raisin exercise, mindful breathing, sitting meditation, sound and thought meditation). Homework assignments (e.g., mindful eating, mindful showering, breathing exercises, compassion meditation) were given at the end of each session, and audio recordings of the meditations were provided for practice. In each subsequent session, participants received verbal feedback on their homework.

ELIGIBILITY:
Inclusion Criteria:

* Those diagnosed with Gestational Diabetes Mellitus,
* Those whose pregnancy is between 24-34 weeks,
* Those who can read and write in Turkish, and those who do not have hearing or speech problems,
* Pregnant women who volunteered to participate in the study.

Exclusion Criteria:

* Those who could not complete the Mindfulness-Based Stress Reduction Program,
* Pregnant women who gave birth while the study was ongoing.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Prenatal Attachment Inventory (PAI) scores | From pre-test (baseline) to 4 weeks post-intervention
  To evaluate the effect of the Mindfulness-Based Stress Reduction Program on prenatal attachment levels in pregnant women with gestational diabetes.
  The four-point Likert-type scale, with each item scored between 1 and 4, consists of a total of 21 items. Participants were asked to select the option most appropriate for them in the inventory as Never (1), Sometimes (2), Often (3), Always (4). The total score that can be obtained from the scale is a minimum of 21 and a maximum of 84 points.
Change in Prenatal Distress Questionnaire (NuPDQ) scores | From pre-test (baseline) to 4 weeks post-intervention
  To evaluate the effect of the Mindfulness-Based Stress Reduction Program on prenatal distress levels in pregnant women with gestational diabetes.
  Participants are asked to mark one of the options listed as Not at all (0), A little (1) and A lot (2) that best suits them regarding whether they are distressed, sad or anxious. The distress score experienced during pregnancy is obtained by adding the scale item scores. The lowest score obtained from the scale is 0, the highest score is 34. As the total score obtained from the scale increases, the level of prenatal distress perceived by pregnant women also increases. The scale has 4 sub-dimensions. They are divided into physical and social changes related to pregnancy, concerns about the baby and birth (Items 1-3-4-6-7-8-10-11-12), concerns about the quality of health care and health status (Items 2-9-17), concerns about the baby's care and life after birth (Items 13-15-16), and financial concerns (Items 5-14).
Change in State-Trait Anxiety Inventory (STAI-S-T) scores | From pre-test (baseline) to 4 weeks post-intervention
  To evaluate the effect of the Mindfulness-Based Stress Reduction Program on state anxiety levels in pregnant women with gestational diabetes.
  STAI-S consists of 20 items; STAI-T, which answers general feelings, consists of 40 items. Both scales are four-point Likert type, and in STAI-S, it is requested to mark the most appropriate option from the options listed as Never (1), A Little (2), A Lot (3), Completely (4), in STAI- Almost Never (1), Sometimes (2), A Lot of Time (3), Almost Always (4). STAI scale shows negative feelings as direct expressions, and positive feelings as reverse expressions. Items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20 in STAI-S Scale and items 26, 27, 30, 33, 36 and 39 in STAI-T Scale are reversed. Direct expressions indicate negative feelings in the individual, and reverse expressions indicate positive feelings in the individual. Scores from both scales vary between 20 and 80.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik Şehir Kadın Doğum Hastanesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No